CLINICAL TRIAL: NCT00101738
Title: Study to Investigate the Clinical Outcomes of Different Regimens of Myfortic® in De Novo Kidney Tx Pts Using Simulect® and Neoral® With or Without Steroids
Brief Title: Freedom Study: Myfortic in Kidney Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Novartis Pharmaceuticals, Novartis
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A2404
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Kidney Transplantation
Keywords: MPA; Kidney Transplantation; Acute rejection; Kidney function
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Myfortic

SUMMARY:
The primary objective of the study is to evaluate that 3 immunosuppressant regimens will have comparable kidney function results in kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 75 years.
* Recipients of first, heart-beating cadaveric, living unrelated or living related non-HLA identical donor kidney transplant, treated with Simulect® and Neoral® as primary immunosuppression.

Exclusion Criteria:

* Second or subsequent kidney transplant or multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any other organ.
* Kidneys from non-heart beating donors or HLA identical living related donors.
* ABO incompatibility against the donor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2003-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Calculated glomerular filtration rate after 12 months treatment

SECONDARY OUTCOMES:
Incidence of death, graft loss, biopsy-proven acute rejection after 3 and 12 months.
Patient and graft survival after 12 months.
Incidence of AEs and SAEs after 3 and 12 months.
Blood pressure, lipids and glucose profiles after 3 and 12 months.
Percentage of patients free of steroids at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (44):
- United States (9):
  - UCSF Kidney Transplant Service, San Francisco, California
  - Livelink, Inc., Tampa, Florida
  - Loyola Medical Center, Maywood, Illinois
  - Indiana U. Medical Center, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - University Hospitals of Cleveland, Division of Nephrology, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Legacy Research & Technology Ctr., Portland, Oregon
  - U. of Wisconsin Hospital Clinics, Madison, Wisconsin
- Argentina (3):
  - Crai Norte, San Martín, Buenos Aires
  - Hospital Cordoba, Córdoba, Córdoba Province
  - Unidad de Transplante Velez Sarsfield, Córdoba, Córdoba Province
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Brazil (2):
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Hipertensao Hospital do Rim e Hipertensao, São Paulo, São Paulo
- Canada (7):
  - Foothills Medical Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Queen II Health and Science Center, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, The Toronto Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Germany (2):
  - Staedt. Krankenhaus Koeln-Merheim, Cologne
  - Klinikum der Johann Wolfgang Geothe-Universitaet, Frankfurt am Main
- Ospedale Consorziale e policlinico-Universita degli Studi, Bari, BA, Italy
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia
- Auckland Hospital, Auckland, Grafton, New Zealand
- Singapore General Hospital, Singapore, Singapore
- Spain (3):
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Central de Asturias, Oviedo, Oviedo
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
- Taiwan (3):
  - Chang-Gung Memorial Hospital-Linko, Taoyuan District, Lin-Ko
  - Taipei Veterans General Hospital, Taipei, ROC
  - National Taiwan University Hospital, Taipei
- United Kingdom (6):
  - Queen Elizabeth Medical Centre, Edgbaston, Birmingham
  - University Hospital of Wales, Heathpark, Cardiff
  - Walsgrave Hospital NHS Trust, Walsgrave on Sowe, Coventry
  - Freeman Hospital, High Heaton, Newcastle Upon Tyne
  - Guy's Hospital, London
  - Nottingham City Hospital, Nottingham